CLINICAL TRIAL: NCT07365202
Title: Osteosynthesis of Fibula Fractures With a Locked Thin Plate: a Single-center Retrospective Series.
Brief Title: Osteosynthesis of Fibula Fractures With a Locked Thin Plate
Acronym: OFFPAV
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC25.0227
Record Dates: First submitted 2026-01-06; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Osteosynthesis of Fibula Fractures With a Locked Thin Plate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ankle fractures represent about 10% of all fractures and are common in both elderly patients with comorbidities and younger polytraumatized individuals. Traditional fibular osteosynthesis uses open plating, which carries up to a 20% complication rate, mainly due to skin issues. These complications are more frequent in patients with diabetes, vascular or neurological disease, obesity, or tobacco/alcohol use, as well as in open fractures or fracture-dislocations. Standard plates can also cause long-term discomfort due to their thickness, often requiring removal.

Recent meta-analyses show that fibular nailing and thin one-third tubular plates result in fewer complications than anatomical plates, while maintaining similar bone-healing rates (97-100%). New thinner locked plates (2.8 mm) have been developed to reduce skin risks and discomfort; biomechanical studies suggest superior strength. Clinical research is needed to confirm their effectiveness and tolerance.

DETAILED DESCRIPTION:
Ankle fractures account for up to 10% of all fractures. They are the third most common fracture site in adults, with nearly 169 cases per 100,000 inhabitants per year . These injuries affect a heterogeneous population, including elderly patients who often have comorbidities as well as younger polytraumatized individuals. Fibular osteosynthesis is traditionally performed by open reduction and internal fixation using plates with screws, either locked or non-locked. The longitudinal approach required for osteosynthesis carries risks, with complication rates reaching up to 20% in some series, the most common being skin complications related to the necessary incision .

The rate of cutaneous complications is associated with age, diabetes, peripheral vascular and neurological diseases, obesity, and alcohol or tobacco use . Moreover, an open injury or a fracture-dislocation further increases this risk. In addition, the plates traditionally used have a certain thickness that can cause long-term discomfort, often requiring hardware removal after bone healing. Recent meta-analyses published show a superiority of fibular nailing-and even simple one-third tubular plates-over so-called "anatomical" plates in terms of complications (patient discomfort, infection, and wound-healing issues), due to the smaller profile of the implants. Bone-healing rates remain comparable across different fixation methods and range from 97% to 100% in recent meta-analyses.

Recently, new implants have been developed to reduce skin risks and discomfort related to implant thickness. These thinner locked plates have a thickness of 2.8 mm (compared with an average of 3.5 mm for competing systems). A recent biomechanical study demonstrated their superior mechanical resistance . A clinical study would be useful to confirm these results in terms of bone healing and tolerance (cutaneous tolerance and implant-related discomfort).

Study designe:Descriptive single-center historico-prospective observational cohort study without a control group

ELIGIBILITY:
Inclusion Criteria:

* Adult patient at the time of injury

  • Patient who underwent surgery with a low-profile plate, including:
  * Isolated lateral malleolar fracture treated with a low-profile anatomical plate
  * Lateral malleolar fracture associated with a bimalleolar injury treated with a low-profile anatomical plate
  * Lateral malleolar fracture associated with a trimalleolar injury treated with a low-profile anatomical plate
  * Lateral malleolar fracture associated with a tibial pilon injury treated with a low-profile anatomical plate
* Standard preoperative radiographs (ankle AP and lateral views)
* Standard postoperative radiographs (ankle AP and lateral views)
* No objection to participation in the study

Exclusion Criteria:

* Individuals deprived of liberty by judicial or administrative decision, or individuals under legal protection
* Patients with dementia preventing the collection of secondary clinical outcome measures (Olerud and Molander score, VAS, EFAS score, EQ-5D-5L)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, all adult patients treated for a lateral malleolus fracture with an anatomically contoured plate, either alone or associated with a bimalleolar, trimalleolar, or tibial pilon injury in the orthopedic and trauma department at Grenoble University Hospital, between 04/01/2025 (the date of first use of the contoured plate) and 1 year post-surgery, may be selected.
  Epidemiological data, preoperative management, fracture types according to the Weber and AO/OTA classifications [12], operative data, as well as radiological data are collected and analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate the clinical of patients treated for fixation of an external malleolus fracture, whether isolated or associated with a bi malleolar, tri malleolar, or tibial pilon injury, using a low profile anatomical plate. | 1 year
  Achieving consolidation without skin complications and without the need for hardware removal.
  * Consolidation is defined as the absence of visible fractures on standard anteroposterior and lateral ankle X-rays at 6 months post-operation.
  * The absence of skin complications is defined as wound healing achieved within the expected theoretical healing period (1 month).
  * The absence of a need for hardware removal is defined as the lack of necessity, one year after surgery, for the patient to have the hardware removed due to discomfort caused by the implant.
Evaluate radiological outcomes of patients treated for fixation of an external malleolus fracture, whether isolated or associated with a bi malleolar, tri malleolar, or tibial pilon injury, using a low profile anatomical plate. | 1 year
  Achieving consolidation without skin complications and without the need for hardware removal.
  * Consolidation is defined as the absence of visible fractures on standard anteroposterior and lateral ankle X-rays at 6 months post-operation.
  * The absence of skin complications is defined as wound healing achieved within the expected theoretical healing period (1 month).
  * The absence of a need for hardware removal is defined as the lack of necessity, one year after surgery, for the patient to have the hardware removed due to discomfort caused by the implant.

SECONDARY OUTCOMES:
Assessment of the quality of radiological reduction | 1 year
  Radiological criteria of McLenann et al (assessment of the quality of radiological reduction)
Evaluation of clinical outcomes: Ankle functional scores | 1 year
  Clinical scores of Olerud and Molander (ankle function score)
Evaluation of clinical outcomes: Pain | 1 year
  Clinical scores of VAS (visual analog scale) , from 0 to 10 (0-10) 0 non pain 10 extreme pain
Evaluation of clinical outcomes: Ankle functional scores | 1 year
  Clinical scores of EFAS (ankle function score)
Evaluation of clinical outcomes: Quality of life | 1 year
  Clinical scores of EQ5D-5L (quality of life)
Evaluation of complications | 1 year
  Complications: re-operation(s), infection, healing disorders, secondary displacement, discomfort from osteosynthesis material, removal of osteosynthesis material

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble Alpes university Hospital, La Tronche, France